CLINICAL TRIAL: NCT05479721
Title: Liver Investigation: Testing Marker Utility in Steatohepatitis (LITMUS): Assessment & Validation of Imaging Modality Performance Across the NAFLD Spectrum in a Prospectively Recruited Cohort
Brief Title: LITMUS Imaging Study
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Newcastle University (Other); University of Nottingham (Other); University of Cambridge (Other); University of Seville (Other); Pinnacle Clinical Research, PLLC (Other); ICAN Nutrition Education and Research (Industry); Assistance Publique - Hôpitaux de Paris (Other); University of Angers (Unknown); University of Palermo (Other); University of Turin, Italy (Other); University Medical Center Mainz (Other); University of Helsinki (Other); University of Bern (Other); Linkoeping University (Other Government); Perspectum (Industry); Antaros Medical (Industry); Resoundant Inc (Unknown); Pfizer (Industry); Novartis (Industry); Takeda (Industry); Intercept Pharmaceuticals (Industry); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: IRAS ID 250344; 18/LO/1953 (Other: NHS Health Research Authority)
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: NAFLD; NASH; NASH - Nonalcoholic Steatohepatitis; Fibrosis, Liver; Steatosis of Liver
Keywords: Liver MultisScan; Magnetic Resonance Elastography; Magnetiic Resonance Imaging; deMILI; diffusion weighted imaging; proton density fat fraction; PDFF; iron corrected T1; cT1; liver stiffness; MRI; MRE; diagnostic study; LITMUS
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis; Fatty Liver; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LITMUS Imaging Study Group: Patients within the European NAFLD Registry who have also consented to participate in the LITMUS Imaging study

SUMMARY:
The LITMUS Imaging Study is a prospectively recruited, observational study of patients with histologically characterised non-alcoholic fatty liver disease (NAFLD). It aims to evaluate the diagnostic performance of imaging biomarkers (ultrasound elastography and magnetic resonance biomarkers) against NAFLD histological scores in a cross-sectional analysis and the natural history of NAFLD in a longitudinal study.

DETAILED DESCRIPTION:
The LITMUS Imaging study is a non-interventional, observational study conducted in parallel to the European NAFLD Registry (NCT04442334), collecting cross-sectional and longitudinal ultrasound elastography and magnetic resonance elastography and imaging data. The LITMUS Imaging study recruits patients with NAFLD who are having a clinically indicated liver biopsy and are already participating in the European NAFLD Registry. Patients in the LITMUS Imaging study have additional imaging assessments at baseline (within 100 days of baseline liver biopsy) and 2 years after baseline (no follow-up biopsy necessary). Imaging assessments include point shear wave elastography, 2D shear wave elastography, MRI scans (Liver Multiscan, deMILI, diffusion weighted imaging, proton density fat fraction, T1 mapping) and MR elastography. Link-anonymised magnetic resonance data are uploaded to a central online portal and analysed centrally by 4 imaging core labs provided by Perspectum (Liver Multiscan), Antaros Medical (MR elastography and DWI), Resoundant (vendor specific PDFF) and University of Seville (deMILI).

ELIGIBILITY:
Inclusion Criteria:

1. Recruited to the European NAFLD Registry
2. Patient had a liver biopsy less than 3 months prior to enrolment into the study or is having a liver biopsy in less than 3 months' time for the assessment of NAFLD.
3. Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

1. Patients that do not speak the language in which the patient information is written will be excluded. Due to the nature of the study, being able to read the information about the study or access to a relevant interpreter is a necessary criterion for participant's safety in regards to MR scanning.
2. Patients judged by the investigator to be unsuitable for inclusion in the study (e.g. where the investigator feels that the participant will not be able to comply with the study procedures)
3. Any contra-indication to Magnetic Resonance Imaging (MRI) (e.g. ferrous metal implants/fragments, implantable cardiac defibrillator or permanent pacemaker, metal clips following neurosurgery, pregnancy, other condition that would make MR scanning unsafe in the opinion of the scanner operator)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known or suspected NAFLD who are undergoing liver biopsy as part of their routine clinical care and are already participating in the European NAFLD Registry
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of imaging biomarkers for severity of liver fibrosis on histology as reference standard | baseline
  sensitivity, specificity, positive predictive value, negative predictive value, area under the receiver operating characteristic curve

SECONDARY OUTCOMES:
Diagnostic accuracy of imaging biomarkers for diagnosis of NASH on histology as reference standard | baseline
  sensitivity, specificity, positive predictive value, negative predictive value, area under the receiver operating characteristic curve
Diagnostic accuracy of imaging biomarkers for histologically assessed fat and iron deposition as reference standard | baseline
  sensitivity, specificity, positive predictive value, negative predictive value, area under the receiver operating characteristic curve
To study the natural history of NAFLD and how this may impact prognosis | evaluation of biomarkers at baseline and after 2 years
  1. Longitudinal correlation of change (δ) in MR and US elastography biomarker values with clinical phenotype data*
  2. Survival analysis for the change (δ) in biomarker values
To evaluate reproducibility and observer dependent variability in reporting of liver imaging biomarkers | evaluation of biomarkers within 30 days
  Statistical correlation of MR and US elastography data obtained from the same patients acquired or analysed on two time points
To identify physiological factors that confound the performance of imaging biomarkers for the assessment of fibrosis | baseline
  Statistical correlation of MR scans and US elastography imaging biomarkers with liver histology parameters (steatosis, iron deposition, inflammation) and other clinical data (demographics, lab results, patient characteristics)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pavlides, MBBS, DPhil, Principal Investigator — University of Oxford
Locations (18):
- Pinnacle Clinical Research, San Antonio, Texas, United States
- Helsinki University Hospital, Helsinki, Finland
- France (2):
  - Le Centre de Recherche Clinique (CRC) du CHU d'Angers, Angers
  - Institut ICAN - Institute of Cardiometabolism And Nutrition Hôpital de la Pitié Salpêtrière, Paris
- Germany (2):
  - UNIVERSITÄTSMEDIZIN der Johannes Gutenberg Universität Mainz, Mainz
  - Universitätsklinikums Würzburg, Würzburg
- Laiko General Hospital of Athens, Athens, Greece
- Italy (2):
  - Università di Palermo, Palermo
  - Department of Medical Sciences University of Torino, Torino
- Spain (3):
  - Vall d'Hebron University Hospital, Barcelona
  - Institute of Biomedicine of Sevilla (IBiS), Virgen del Rocío University Hospital, Seville
  - HU Clínico de Valladolid, Valladolid
- Linköping University Hospital, Linköping, Sweden
- Inselspital, University Hospital, Bern, Switzerland
- United Kingdom (4):
  - Addenbrookes Hospital, Cambridge
  - The Newcastle Upon Tyne Hospitals Nhs Foundation Trust, Newcastle upon Tyne
  - Queens Medical Centre, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pavlides M, Mozes FE, Akhtar S, Wonders K, Cobbold J, Tunnicliffe EM, Allison M, Godfrey EM, Aithal GP, Francis S, Romero-Gomez M, Castell J, Fernandez-Lizaranzu I, Aller R, Gonzalez RS, Agustin S, Pericas JM, Boursier J, Aube C, Ratziu V, Wagner M, Petta S, Antonucci M, Bugianesi E, Faletti R, Miele L, Geier A, Schattenberg JM, Tilman E, Ekstedt M, Lundberg P, Berzigotti A, Huber AT, Papatheodoridis G, Yki-Jarvinen H, Porthan K, Schneider MJ, Hockings P, Shumbayawonda E, Banerjee R, Pepin K, Kalutkiewicz M, Ehman RL, Trylesinksi A, Coxson HO; LITMUS Consortium Investigators; Martic M, Yunis C, Tuthill T, Bossuyt PM, Anstee QM, Neubauer S, Harrison S. Liver Investigation: Testing Marker Utility in Steatohepatitis (LITMUS): Assessment & validation of imaging modality performance across the NAFLD spectrum in a prospectively recruited cohort study (the LITMUS imaging study): Study protocol. Contemp Clin Trials. 2023 Nov;134:107352. doi: 10.1016/j.cct.2023.107352. Epub 2023 Oct 4. PMID 37802221